CLINICAL TRIAL: NCT00407706
Title: Breast Cancer- Early Detection of Cancer Disease and Pre-Cancer Disease, and in Women That Are at High Risk for Developing Breast Cancer by Identifying Lymphocytes Previously Exposed to Specific Cancer Antigen.
Brief Title: Using Test of SCM for Detection Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Other Study IDs: HP 6-218 S
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Malignant Breast Cancer, Benign Breast Lesions
Keywords: Breast Cancer, FACS, SCM, Malignant, Benign, Lymphocytes
MeSH Terms: conditions — Breast Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: blood test

SUMMARY:
In our previous research, we have shown that women that have breast cancer have a population of lymphocytes that recognizes specific antigen and there cytoplasmic matrix goes through physical change a short time after exposure in vitro to the same antigen. This change can be measured by polarization changes of fluorescent light emitted by FDA (fluorescein diacetate) labeled cells. Further test that we performed showed that those differences are also shown in a benign situation that known as indicator for a high risk for developing breast cancer within 10-15 years. The incidence of the expression of these lymphocytes correlates with the histopathological picture as it is related in high risk for the developing the disease.

In this work we will expand the scope of the procedure to early detection of the cancerous process in breast lesions by Fitzgibbon's risk categories for the development invasive carcinoma of the breast. In the proposed work we intend to use specific antigen MUC1 for breast cancer. This study is a continuation of our published work in the "The Breast "

ELIGIBILITY:
Inclusion Criteria:

Women carrying benign breast lesions will be further divided and analyzed according to the Fitzgibbon's risk categories for invasive cancer risk (4). The Fitzgibbon's categories are:

1. No increased risk group including adenosis (other than sclerotic), duct ectasia fibroadenoma without complex features,
2. slightly increased risk group (1.5-20 times) which includes fibroadenoma with complex features, moderate or florid hyperplasia without atypia, sclerosing adenosis,
3. moderately increased risk group (4.0-5.0 times) includes atypical ductal and lobular hyperplasia and
4. markedly increased risk group (8.0-10.0 times) which includes ductal and lobular carcinomas In Situ Following the blood collection, detailed relevant clinical information of the patient will be registered in a case record form.

The data will include: age, country of birth, last menstrual period, lactation, number of children, age at first full-term pregnancy, age at onset of menopause, family history, medication, mammography findings, FNA results, tumor size, histological findings, biopsies, disease staging, and other relevant clinical information.

Exclusion Criteria:

1. pregnancy,
2. experiencing menstruation, or
3. under hormonal or drug treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180
Dates: Start 2006-12; Study Completion 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Amram Hadari, MD, Principal Investigator — Surgery Department
Locations (1):
- Surgery Department, Safed, Israel

REFERENCES:
- [Background] Klein O, Lin S, Embon O, Sazbon A, Zidan J, Kook AI. An approach for high sensitivity detection of prostate cancer by analysis of changes in structuredness of the cytoplasmic matrix of lymphocytes specifically induced by PSA-ACT. J Urol. 1999 Jun;161(6):1994-6. PMID 10332488
- [Background] Klein O, Linn S, Hadari A, Davidson C, Eitan A, Zidan J, Kook AI. An approach for high sensitivity detection of breast cancer by analysis of changes in structure of the cytoplasmic matrix of lymphocytes specifically induced by a specific breast tumour antigen (MUC-l/SEC). Breast. 2002 Apr;11(2):137-43. doi: 10.1054/brst.2001.0315. PMID 14965660
- [Background] Fitzgibbons PL, Henson DE, Hutter RV. Benign breast changes and the risk for subsequent breast cancer: an update of the 1985 consensus statement. Cancer Committee of the College of American Pathologists. Arch Pathol Lab Med. 1998 Dec;122(12):1053-5. PMID 9870852
- [Background] Smorodinsky N, Weiss M, Hartmann ML, Baruch A, Harness E, Yaakobovitz M, Keydar I, Wreschner DH. Detection of a secreted MUC1/SEC protein by MUC1 isoform specific monoclonal antibodies. Biochem Biophys Res Commun. 1996 Nov 1;228(1):115-21. doi: 10.1006/bbrc.1996.1625. PMID 8912645
- [Background] Karanikas V, Hwang LA, Pearson J, Ong CS, Apostolopoulos V, Vaughan H, Xing PX, Jamieson G, Pietersz G, Tait B, Broadbent R, Thynne G, McKenzie IF. Antibody and T cell responses of patients with adenocarcinoma immunized with mannan-MUC1 fusion protein. J Clin Invest. 1997 Dec 1;100(11):2783-92. doi: 10.1172/JCI119825. PMID 9389743
- [Background] Hiltbold EM, Ciborowski P, Finn OJ. Naturally processed class II epitope from the tumor antigen MUC1 primes human CD4+ T cells. Cancer Res. 1998 Nov 15;58(22):5066-70. PMID 9823312
- [Background] Kelly JM, Darcy PK, Markby JL, Godfrey DI, Takeda K, Yagita H, Smyth MJ. Induction of tumor-specific T cell memory by NK cell-mediated tumor rejection. Nat Immunol. 2002 Jan;3(1):83-90. doi: 10.1038/ni746. Epub 2001 Dec 17. PMID 11743585
- [Result] Klein O, Linn S, Davidson C, Hadary A, Shukha A, Zidan J, Eitan A, Kook AI. Early detection of malignant process in benign lesions of breast tumor by measurements of changes in structuredness of cytoplasmic matrix in circulating lymphocytes (SCM test) reinduced in vitro by specific tumor antigen. Breast. 2002 Dec;11(6):478-83. doi: 10.1054/brst.2002.0477. PMID 14965713